CLINICAL TRIAL: NCT01525082
Title: A Phase 2 Study of Capecitabine, Temozolomide, and Bevacizumab for Metastatic or Unresectable Pancreatic Neuroendocrine Tumors
Brief Title: Capecitabine, Temozolomide, and Bevacizumab for Metastatic or Unresectable Pancreatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaheen Shagufta (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Shaheen Shagufta, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-22412; NCI-2011-03497 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SU-10282011-8571 (Other: Stanford University); NET0012 (Other: OnCore); END0012 (Other: superceded OnCore); 4593 (Other: superceded IRB number)
Record Dates: First submitted 2012-01-10; First posted 2012-02-02 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Gastrinoma; Glucagonoma; Insulinoma; Pancreatic Polypeptide Tumor; Recurrent Islet Cell Carcinoma; Recurrent Pancreatic Cancer; Somatostatinoma; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Carcinoma, Islet Cell; Pancreatic Neoplasms; Somatostatinoma | interventions — Capecitabine; Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bevacizumab + Capecitabine + Temozolomide (Experimental): Cycles repeat every 28 days until disease progression, unacceptable toxicity, or withdrawal.
  Interventions: Drug: Capecitabine; Drug: Temozolomide; Biological: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine — Capecitabine by mouth twice daily on Days 1 to 14
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Drug: Temozolomide — Temozolomide by mouth daily on Days 10 to 14
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Biological: Bevacizumab — Bevacizumab IV over 30 to 90 minutes on Days 1 & 15
  Other Names: Avastin; anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; rhuMAb VEGF

SUMMARY:
The purpose of this research is to evaluate the effectiveness and safety of a combination of capecitabine, temozolomide and bevacizumab in the treatment of advanced pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* Estimate if the combination of capecitabine and temozolomide with bevacizumab for metastatic or unresectable neuroendocrine tumors will improve response rate (RR) by 62% over historical controls (null RR of 40% to true RR 65%).
* Assess the toxicities using Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

SECONDARY OBJECTIVES:

* Evaluate progression-free survival (PFS) and overall survival (OS) using Kaplan-Meier analysis.
* Assess O6-methyl guanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) at baseline by central pathology (path) review.
* Assess serum hormone marker levels.
* Evaluate computed tomography (CT) Perfusion as a tool to predict early therapeutic response. (Optional)
* Bank serum for future correlative analyses.

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30 to 90 minutes on days 1 and 15, capecitabine orally (PO) twice daily (BID) on days 1 to 14, and temozolomide PO once daily (QD) on days 10 to 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity, with assessment for treatment effect every 3 cycles.

After completion of study treatment, patients are followed up patients are followed long-term for survival.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically-confirmed pancreatic neuroendocrine tumors that are moderately- or well-differentiated
* Metastatic or unresectable disease
* If prior surgical resection > 5 years before the development of metastatic disease, a separate (recent) histological or cytological confirmation of metastatic disease is required
* If there is substantial clinical ambiguity regarding the nature or source of apparent metastases, clinicians should consider biopsy of lesions to establish diagnosis of metastatic disease
* The site of previous radiotherapy, if the only site of disease, has evidence of progressive disease
* If prior sunitinib and everolimus has been administered, a 2-week wash-out period is required prior to 1st dose on this study
* If prior liver-directed therapies (ie, chemoembolization, radioembolization), target lesions in the liver have demonstrated growth since the liver-directed treatment
* If prior peptide receptor radionuclide therapy (PRRT), target lesions in the liver have demonstrated growth since the liver-directed treatment
* Low-dose aspirin (≤ 325 mg/d) may be continued in subjects at higher risk for arterial thromboembolic disease.
* Primary or metastatic tumor lesion measurable in at least 1 dimension, within 4 weeks prior to entry of study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* ≥ 18 years of age.
* Laboratory values as follows, ≤ 2 weeks prior to randomization:
* Absolute neutrophil count (ANC) ≥ 1.5 x 10e9/L (≥ 1500/mm³)
* Platelets (PLT) ≥ 100 x 10e9/L (≥ 100,000/mm³)
* Hemoglobin (Hgb) ≥ 9 g/dL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
* Serum bilirubin ≤ 1.5 x ULN
* Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) ≤ 3.0 x ULN (≤ 5.0 x ULN if liver metastases present). Note: endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous stenting may be used to normalize the liver function tests
* Urine dipstick or urinalysis for protein, value must be 0, trace, or 1+ protein to enroll. EXCEPTION: if ≥ 2+ must check 24-hour urine protein and must be < 1 g
* Life expectancy ≥ 12 weeks
* Ability to give written informed consent according to local guidelines
* If any prior therapy-related toxicities, must have recovered from all

EXCLUSION CRITERIA Disease-Specific Exclusions

* Prior bevacizumab; fluoropyrimidines (eg, capecitabine or 5-fluorouracil, 5FU); or temozolomide
* Poorly-differentiated or high-grade pancreatic neuroendocrine tumors
* Prior full field radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to enrollment
* Diagnosis of another malignancy, unless > 3 years earlier and has been disease-free for > 6 months following the completion of curative intent therapy, specific eligibility exceptions as follows:
* Curatively-resected non-melanomatous skin cancer
* Curatively-treated cervical carcinoma in situ
* Organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values, if hormonal therapy has been initiated or a radical prostatectomy has been performed
* Other primary solid tumor curatively treated with no known active disease present and no treatment administered for > 3 years
* Concurrent use of other investigational agents and patients who have received investigational drugs ≤ 4 weeks prior to enrollment
* Known hypersensitivity to capecitabine, temozolomide, or any component of the formulation
* Known deficiency of dihydropyrimidine dehydrogenase Bevacizumab-specific Exclusions
* Inadequately-controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known central nervous system (CNS) metastases
* Significant vascular disease (eg, aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (≥ ½ teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Known hypersensitivity to any component of bevacizumab General Medical Exclusions
* Inability to comply with study and/or follow-up procedures
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study
* Pregnant or lactating/breast feeding
* Lack of effective contraception men or women of child-bearing potential
* Uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Known history of HIV, HBV, or HCV
* Current, ongoing treatment with full-dose warfarin. However, patients may be on stable doses of a low-molecular weight heparin are allowed [eg, (enoxaparin (Lovenox)].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2018-01 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Shagufta, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Capecitabine + Temozolomide: Cycles repeat every 28 days until disease progression, unacceptable toxicity, or withdrawal. Assessments for treatment effect are after every 3 cycles of treatment.
  * Capecitabine: Capecitabine by mouth twice daily on Days 1 to 14
  * Temozolomide: Temozolomide by mouth daily on Days 10 to 14
  * Bevacizumab: Bevacizumab IV over 30 to 90 minutes on Days 1 & 15
Period: Overall Study
Arm/Group | Bevacizumab + Capecitabine + Temozolomide
Started | 20
Completed (Completion defined as assessment for clinical response after 3 cycles of treatment.) | 19
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + Capecitabine + Temozolomide
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response (RR)
Description: Tumor response to treatment with the combination of capecitabine & temozolomide plus bevacizumab in patients with metastatic or unresectable pancreatic neuroendocrine tumors was assessed per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions. Response is defined as:
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
  The outcome is reported as the number of participants who between 3 and 18 months after treatment initiation achieve CR, PR, or clinical response (PR + CR), each a number without dispersion.
Time Frame: 18 months
Population: Not all participants were evaluable for response to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + Capecitabine + Temozolomide
Number analyzed (Participants) | 19
Participants
  Overall response (OR) | 9
  Complete Response (CR) | 0
  Partial Response (PR) | 9
  Stable Disease (SD) | 9
  Progressive disease (PD) | 1

2. Secondary Outcome: Treatment-related Toxicity
Description: Patients will be monitored for hematologic (blood and lymphatic), gastrointestinal (stomach and gut), renal (kidney), liver (metabolic), neurological, and systemic (constitutional) toxicities (treatment-related adverse events). Toxicity events occurring during treatment will be tabulated for each indicated organ system, and listed separated for serious and non-serious events, with the toxicity attribution indicated. The outcome is reported as the number of events, a number without dispersion.
Time Frame: 18 months
Measure: Number; unit: Toxicities (treatment-related events)
Groups:
- Bevacizumab: Toxicities attributed to bevacizumab
- Capecitabine: Toxicities attributed to capecitabine
- Temozolomide: Toxicities attributed to temozolomide
Arm/Group | Bevacizumab | Capecitabine | Temozolomide
Number analyzed (Participants) | 20 | 20 | 20
Toxicities (treatment-related events)
  Serious blood or lymphatic | 1 | 0 | 0
  Serious gastrointestinal | 1 | 0 | 0
  Serious kidney | 1 | 0 | 0
  Serious nervous system | 1 | 0 | 0
  Non-serious blood or lymphatic | 1 | 5 | 8
  Non-serious gastrointestinal | 34 | 119 | 77
  Non-serious systemic | 11 | 59 | 56
  Non-serious kidney | 69 | 0 | 0
  Non-serious metabolism | 3 | 15 | 12
  Non-serious nervous system | 12 | 16 | 12

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) means the length of time that participants survive without disease (tumor) progression, and was assessed using Kaplan-Meier analysis. The outcome is given as the mean in months with standard error of the mean.
Time Frame: 82 months
Population: Participants lost to follow-up are not included. The data are final. Participants are not being followed for additional data or analysis.
Measure: Mean (Standard Error); unit: months
Arm/Group | Bevacizumab + Capecitabine + Temozolomide
Number analyzed (Participants) | 20
months | 25.2 (3.3)

4. Secondary Outcome: Overall Survival (OS)
Description: Time from the date of enrollment to the date of death due to any cause or the last date the patient was known to be alive (censored observation) at the date of data cutoff for the final analysis. The results will be reported as median in months
  The length of overall survival (OS) of participants was assessed by Kaplan-Meier analysis. The outcome is given as the median in months with full range.
Time Frame: 82 mo
Population: The data are final. Participants are not being followed for additional data or analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab + Capecitabine + Temozolomide
Number analyzed (Participants) | 20
months | 49.8 [2.3 to 81.9]

5. Secondary Outcome: O6-methylguanine DNA Methyltransferase (MGMT) Status by Immunohistochemistry (IHC)
Description: O6-alkylguanine DNA alkyltransferase is a protein that in humans is encoded by the gene "O6-methylguanine DNA methyltransferase" (MGMT). Deficiency of the gene product, ie, the protein, is refereed to as "MGMT deficiency," and is thought to be predictive of response to temozolomide and is more often associated with pancreatic NETs.
  MGMT status in pre-treatment biopsy specimens was to be assessed by immuno-histochemistry (IHC), and associated to best clinical response. The outcome is reported by the the number of patients that were IHC-positive (MGMT detected) or IHC-negative (MGMT not detected), and by best clinical response [ie, complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD)]. The outcome is reported as a number without dispersion.
Time Frame: 18 months
Population: For some participants, tissue was not collected, insufficient tissue was collected, or the tissue analysis failed (no result).
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Capecitabine + Temozolomide
Number analyzed (Participants) | 11
participants
  IHC-positive and CR | 0
  IHC-positive and PR | 2
  IHC-positive and SD | 2
  IHC-positive and PD | 1
  IHC-negative and CR | 0
  IHC-negative and PR | 4
  IHC-negative and SD | 2
  IHC-negative and PD | 0

6. Secondary Outcome: O6-methylguanine DNA Methyltransferase (MGMT) by Promoter Methylation
Description: O6-alkylguanine DNA alkyltransferase is a protein that in humans is encoded by the gene "O6-methylguanine DNA methyltransferase" (MGMT). Deficiency of the gene product, ie, the protein, is refered to as "MGMT deficiency," and is thought to be predictive of response to temozolomide and is more often associated with pancreatic NETs.
  MGMT status in pre-treatment biopsy specimens was to be assessed by extent of genetic promoter methylation (an analysis of DNA), and correlated to subject survival.
  MGMT status in pre-treatment biopsy specimens was to be assessed by promoter methylation assessment (PM), and associated to best clinical response. The outcome is reported by the the number of patients that were PM-positive (MGMT detected) or PM-negative (MGMT not detected), and by best clinical response [ie, complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD)]. The outcome is reported as a number without dispersion.
Time Frame: 18 months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Capecitabine + Temozolomide
Number analyzed (Participants) | 11
participants
  PM-positive and CR | 0
  PM-positive and PR | 1
  PM-positive and SD | 0
  PM-positive and PD | 0
  PM-negative and CR | 0
  PM-negative and PR | 4
  PM-negative and SD | 5
  PM-negative and PD | 1

ADVERSE EVENTS:
Time Frame: 18 months
Description: This study is a single cohort of one combination treatment. Overall adverse events were collected and reported for the single cohort. No attempt will be made to conduct a retrospective analysis attributing adverse events per an analytical plan not defined in the protocol.
Groups:
- Bevacizumab + Capecitabine + Temozolomide: Cycles repeat every 28 days until disease progression, unacceptable toxicity, or withdrawal.
  * Capecitabine: Capecitabine by mouth twice daily on Days 1 to 14
  * Temozolomide: Temozolomide by mouth daily on Days 10 to 14
  * Bevacizumab: Bevacizumab IV over 30 to 90 minutes on Days 1 & 15
Arm/Group | Bevacizumab + Capecitabine + Temozolomide
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 20/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Capecitabine + Temozolomide (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Capecitabine + Temozolomide (N=20)
Anemia (Blood and lymphatic system disorders) | 7 (11)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (3)
Palpitations (Cardiac disorders) | 3 (5)
Chest pain (Cardiac disorders) | 3 (6)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Watering eyes (Eye disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (36)
Vomiting (Gastrointestinal disorders) | 9 (19)
Constipation (Gastrointestinal disorders) | 15 (30)
Diarrhea (Gastrointestinal disorders) | 11 (39)
Bloating (Gastrointestinal disorders) | 5 (8)
Oral hemorrhage (Gastrointestinal disorders) | 8 (18)
Hemorrhoids (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 5 (9)
Abdominal pain (Gastrointestinal disorders) | 13 (30)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 (7)
Oral pain (Gastrointestinal disorders) | 4 (6)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2)
Lip pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (4)
Toothache (Gastrointestinal disorders) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 1 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (2)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 16 (57)
Pain (General disorders) | 5 (44)
Edema limbs (General disorders) | 7 (11)
General disorders and administration site conditions - Other (General disorders) | 2 (3)
Fever (General disorders) | 4 (6)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (4)
Injection site reaction (General disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 5 (5)
Paronychia (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (3)
Alanine aminotransferase increased (Investigations) | 13 (37)
Aspartate aminotransferase increased (Investigations) | 12 (34)
Platelet count decreased (Investigations) | 11 (32)
Lymphocyte count decreased (Investigations) | 12 (38)
Blood bilirubin increased (Investigations) | 5 (30)
Creatinine increased (Investigations) | 10 (27)
Alkaline phosphatase increased (Investigations) | 7 (17)
White blood cell decreased (Investigations) | 6 (12)
Neutrophil count decreased (Investigations) | 5 (12)
Weight loss (Investigations) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Weight gain (Investigations) | 4 (6)
Lymphocyte count increased (Investigations) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 5 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (10)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (17)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (61)
Hypokalemia (Metabolism and nutrition disorders) | 3 (9)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 13 (30)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (6)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (17)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Headache (Nervous system disorders) | 10 (22)
Concentration impairment (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (6)
Sinus pain (Nervous system disorders) | 3 (8)
Memory impairment (Nervous system disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (2)
Depression (Psychiatric disorders) | 4 (5)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (3)
Proteinuria (Renal and urinary disorders) | 13 (53)
Hematuria (Renal and urinary disorders) | 9 (20)
Urinary frequency (Renal and urinary disorders) | 1 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (30)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 (12)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 (28)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 7 (8)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 15 (69)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT01525082/Prot_SAP_000.pdf